CLINICAL TRIAL: NCT00733616
Title: Phase II Study of Adjusted-dose Docetaxel-oxaliplatin-capecitabine in Patients With Advanced Gastric Adenocarcinoma and Intermediate General Status.
Brief Title: Efficacy and Safety Study of Combination Therapy With Docetaxel-oxaliplatin-capecitabine in Patients With Advanced Gastric Adenocarcinoma and Intermediate General Status
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Sanofi (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-08-02; EudraCT Nº: 2008-001825-32
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Gastric Cancer
Keywords: advanced gastric adenocarcinoma; docetaxel; oxaliplatin; capecitabine; intermediate general status
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: DOX: Docetaxel, oxaliplatin, Capecitabine

INTERVENTIONS:
Drug: DOX: Docetaxel, oxaliplatin, Capecitabine — * Docetaxel 40 mg/m2, iv infusion 60 minutes, day 1
  * Oxaliplatin 80 mg/m2, iv infusion 120 minutes, day 1
  * Capecitabine 625 mg/m2, bid, oral, continuous
    6 cycles, every 3 weeks
  Capecitabine will be given same dose (625mg/m2/bid) continuous in case no toxicity (no dose adjustment)

SUMMARY:
The purpose of the study is to determine efficacy and safety of combination therapy with adjusted-dose docetaxel-oxaliplatin-capecitabine in patients with advanced gastric adenocarcinoma and intermediate general status.(defined as ECOG 2 or weight loss 10-25% or older that 70 years and no comorbidities nor functional dependency nor geriatric syndrome)

ELIGIBILITY:
Inclusion Criteria:

1. informed consent signed
2. Histological or cytological adenocarcinoma confirmation carcinoma on the esophago-gastric union or stomach (type I, II and III Siervent) metastatic or relapsed
3. measurable disease (following RECIST criteria)
4. older or equal 70 years old
5. Intermediate general status defined as at least one of the following characteristics: performance status (ECOG) = 2, weight loss ponderada between 10 and 25% in the last 3 months
6. life expectancy superior to 12 weeks
7. adequate hematological function: Neutrophils ≥1.50x109, platelets ≥100x109, Hemoglobin ≥10 g/dl
8. adequate liver function: Liver function (total bilirubine < 2 NV; GOT y GPT <3 NV (< 5 NV in case of liver metastasis; Alkaline phosphatase <3 NV ))
9. Adequate renal function: renal function (Creatinine clearance > 50mL/min), based on Cockroff - Gault. In case Creatinine clearance is < 50 ml/min, a test in urine will be done in 24 hours and if the value is > 50 ml/min, the patient could be eligible for the study
10. Potential fertile women negative pregnancy test in serum or urine, 10 days prior the first study dose given
11. Use an adequate contraceptive method (postmenopausal women should be amenorrheic at least 12 months previous the study to be considered as not potentially fertile (VN:upper limit on normal laboratory values)

Exclusion Criteria:

1. non measurable lesion as only disease evidence
2. previous chemotherapy treatment for advance disease. It wont´t be consider as exclusion criteria if chemo or radiotherapy has been given for localized disease and finished more than 1 year ago. In caso os only measurable disease in the radiated area, progressive disease has to be documented previous to the inclusion
3. functional dependency
4. hypersensitivity to Docetaxel, oxaliplatin or capecitabine
5. previous serious adverse events or unexpected to fluoropirimidin treatment and /or patients with proved deficit in dehidropirimidin deshidrogenase (DPD)
6. patients classified as "weak or fragile"

   1. dependency on one or more of the daily activities following the daily activity scale from Katz
   2. three or more comorbitities of the following: congestive cardiac insufficiency, cardiac valvulopathy, coronaripathia, chronic pulmonary disease (obstructive or restrictive), cerebrovascular disease, diabetes, concomitant neoplasms, collagen vascular disease, chronic hetopathy and incapacitate arthritis
   3. presence of geriatric syndromes: moderate-severe dementia, stress delirium (urinary respiratory infection); moderate-severe depression that interfere in the habitual daily life; frequent falls (3 or more monthly); be disattended; urinary incontinence, without stress, infection, diuretics or prostatic hyperplasia; fecal incontinence without diarrhea or laxative; osteoporotic fracture of long bone or vertebral squash
7. Cardiac concomitant present:

   1. Symptomatic auriculoventricular arrhythmia history, and /or
   2. Congestive cardiac insufficiency non controlled by drugs, and / or
   3. Myocardial infarct 12 months previous the inclusion, and /or
   4. Symptomatic ischemic cardiopathy
8. active infectious process ((leukocytes superior to 12 x 109/l or fever upper to 38º, it is required thorax X:ray, hemoculture and urine culture 5 days previous to the inclusion)
9. severe or bad controlled concomitant disease
10. neoplastic history (except skin basocellular or in-situ cervical carcinoma properly treated) in the last 5 years
11. patients with any other medical or surgical important problem that, in the investigator opinion, could not allow to follow the treatment
12. not able to fulfill the protocol and follow-up
13. being involve in any investigational trial with any drug within 4 weeks prior the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
objective response rate | 2008-2011

SECONDARY OUTCOMES:
adverse events | 2008-2011
Progression free survival (PFS), time to treatment failure (TTF), overall survival and dose intensity | 2008-2011

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Rivera, MD; phD, Study Chair — Hospital Marques de Valdecilla. Santander. Spain
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy, Madrid, Spain

REFERENCES:
- [Derived] Rivera F, Massuti B, Salcedo M, Sastre J, Martinez Galan J, Valladares-Ayerbes M, Serrano R, Garcia de Paredes ML, Manzano JL, Galan M, Alsina M, Yuste Izquierdo AL, Lopez C, Diaz-Rubio E, Conde V, Reboredo M, Cano MT, Pachon V, Aranda E. Phase II trial of miniDOX (reduced dose docetaxel-oxaliplatin-capecitabine) in "suboptimal" patients with advanced gastric cancer (AGC). TTD 08-02. Cancer Chemother Pharmacol. 2015 Feb;75(2):319-24. doi: 10.1007/s00280-014-2641-3. Epub 2014 Dec 10. PMID 25491381